CLINICAL TRIAL: NCT03326843
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Avatrombopag for the Treatment of Subjects With Thrombocytopenia Scheduled for a Surgical Procedure
Brief Title: Avatrombopag for the Treatment of Thrombocytopenia in Adults Scheduled for a Surgical Procedure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to enrollment challenges.
Sponsor: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA-PST-320
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2018-05

CONDITIONS: Thrombocytopenia
Keywords: low platelet count; ITP
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avatrombopag 60 mg (Experimental): Open-label: oral avatrombopag
  Interventions: Drug: Avatrombopag 60 mg

INTERVENTIONS:
Drug: Avatrombopag 60 mg — Oral avatrombopag administered once daily for 5 days prior to procedure.

SUMMARY:
Phase 3b open-label, multicenter study to evaluate the safety and efficacy of avatrombopag in subjects with thrombocytopenia scheduled for operations to critical sites or operations with a high risk of bleeding.

DETAILED DESCRIPTION:
Subjects will receive oral avatrombopag once daily for 5 days beginning on Day 1, followed by a wait period prior to the procedure, which will occur on Day 10 to 13. The Follow-up Period will include 2 visits; 7 days post-procedure and 30 days after last dose.

ELIGIBILITY:
Inclusion Criteria:

* Men and women greater than or equal to 18 years of age;
* A mean baseline platelet count between:

  * 50 × 10^9/L and <100 × 10^9/L for non-chronic liver disease participants
  * 50 × 10^9/L and <75 × 10^9/L for participants with chronic liver disease;
* Participant is scheduled to undergo operations to critical sites (eg, eye surgery, neurosurgery) or operations with a high risk of bleeding (eg, major abdominal surgery), or, in the opinion of the Investigator, would otherwise require a pre-operative platelet transfusion to prevent bleeding

Exclusion Criteria:

* Participant with a history of arterial or venous thrombosis within 6 months of baseline;
* Participant with known portal vein blood flow velocity rate <10 cm/second or previous portal vein thrombosis within 6 months of baseline;
* Participant plans to have a platelet transfusion or plans to receive blood products containing platelets within 7 days of the Baseline Visit;
* Use of erythropoietin-stimulating agents;
* Participant has a known medical history of genetic prothrombotic syndromes; or
* Participant has abnormal hemoglobin levels or prothrombin time/international normalized ratio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Dova Site, Little Rock, Arkansas
  - Dova Site, Coronado, California
  - Dova Site, Aurora, Colorado
  - Dova Site, Jacksonville, Florida
  - Dova Site, Miami, Florida
  - Dova Site, Pensacola, Florida
  - Dova Site, Sarasota, Florida
  - Dova Site, Tamarac, Florida
  - Dova Site, Tampa, Florida
  - Dova Site, New Orleans, Louisiana
  - Dova Site, Baltimore, Maryland
  - Dova Site, Boston, Massachusetts
  - Dova Site, Detroit, Michigan
  - Dova Site, Springfield, Missouri
  - Dova Site, St Louis, Missouri
  - Dova Site, Reno, Nevada
  - Dova Site, Englewood, New Jersey
  - Dova Site, Buffalo, New York
  - Dova Site, Durham, North Carolina
  - Dova Site, Winston-Salem, North Carolina
  - Dova Site, Toledo, Ohio
  - Dova Site, Bethlehem, Pennsylvania
  - Dova Site, Austin, Texas
  - Dova Site, Newport News, Virginia
  - Dova Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avatrombopag 60 mg
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avatrombopag 60 mg
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 66 [51 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Platelet Counts [Mean (Full Range); unit: 10^9 platelets/L] | 68 [64 to 73]

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Efficacy of Avatrombopag in Increasing Platelet Counts in Subjects With Thrombocytopenia Scheduled for Operations
Description: Proportion of subjects that achieve a platelet count >100 x 10^9 platelets/L on procedure day
Time Frame: Baseline to 10-13 days
Measure: Number; unit: proportion of total participants
Arm/Group | Avatrombopag 60 mg
Number analyzed (Participants) | 4
proportion of total participants | 0.75

2. Secondary Outcome: Evaluate Safety of Avatrombopag: Incidence of Treatment Emergent Adverse Events
Description: Incidence of treatment emergent adverse events
Time Frame: Up to 35 days
Population: Study was early terminated due to low enrollment
Arm/Group | Avatrombopag 60 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the time of consent through study follow up visit, up to 35 days.
Arm/Group | Avatrombopag 60 mg
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avatrombopag 60 mg (N=4)
Influenza (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following a multicenter publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Institution shall remove from the proposed publication any information that is considered confidential other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03326843/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03326843/SAP_001.pdf